CLINICAL TRIAL: NCT06095999
Title: Perfect Fit: A Mixed-methods Evaluation of a Virtual Coach Using Personalized Real-time Feedback to Promote Smoking Cessation and Physical Activity
Brief Title: Perfect Fit: Evaluation of a Virtual Coach for Smoking Cessation and Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, aversluis, Dr. (Assistant professor), Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: N23.045 METC-LDD; 628.011.211 (Other Grant/Funding Number: NWO program Commit2Data - Big Data & Health)
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-03

CONDITIONS: Smoking; Low Physical Activity Level
Keywords: Smoking; Smoking Cessation; Physical Activity; Virtual Coach; Chatbot; Relapse Prevention; eHealth; low physical activity
MeSH Terms: conditions — Smoking; Smoking Cessation; Motor Activity

STUDY DESIGN:
Intervention Model Description: A mixed-method single-arm pre-post intervention study will be used. Baseline questionnaires (T0) measure demographic, PA and smoking-characteristics. Post-intervention questionnaires (T1) measuring feasibility of the study and Perfect Fit intervention, acceptability of the Perfect Fit intervention and virtual coach, and preliminary effectiveness of the Perfect Fit intervention will be administered 16 weeks after the start of the intervention (i.e., expected end of intervention). Participants who consent to take part in the semi-structured individual interview will be invited for this interview also around 16 weeks after the start of the intervention. Finally, follow-up questionnaires measuring preliminary effectiveness of the Perfect Fit intervention will be administered 24 (T2), 40 (T3), and 64 (T4) weeks after the start of the intervention (i.e., respectively 2, 6 and 12 months after expected end of the intervention).
Masking Description: N/A due to single-arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 'Perfect Fit' virtual coaching intervention (Experimental): Due to the single-arm design, all participants will receive the Perfect Fit intervention, a personalized eHealth intervention that supports them to stop smoking and increase their PA using a virtual coach (i.e., chatbot).
  Interventions: Behavioral: Perfect Fit intervention: virtual coaching intervention to quit smoking and increase physical activity

INTERVENTIONS:
Behavioral: Perfect Fit intervention: virtual coaching intervention to quit smoking and increase physical activity — The intervention, delivered through a virtual coach, has a personalized duration and intensity, but will last on average 16 weeks. The intervention has three phases: preparation, execution (including [re]lapse) and closing. By having chat conversations with the Perfect Fit virtual coach (using the mobile application 'NiceDay'), the user will be guided through the different phases of the intervention. In each phase, the user has chat conversations with the virtual coach (e.g. about goal setting, weekly reflection) and, in addition, receives exercises and educational video material to support smoking cessation and PA promotion. Additionally, a smartwatch is used to objectively assess PA. It allows participants to monitor their PA and the data (on the number of steps) is used to give automatic, personalized PA advice to the user.

SUMMARY:
The leading cause of disease burden across the globe is cardiovascular disease (CVD). Important modifiable behavioral CVD risk factors include, amongst others, smoking and low physical activity (PA). Individuals with a low socioeconomic position (SEP) often have a less favorable profile of risk factors, resulting in a higher disease burden and premature death. There is a need for cost-effective multi-behavior interventions that target one or more risk factors. eHealth applications are increasingly being used to offer behavior change interventions. Potential benefits include accessibility, scalability, cost-effectiveness, and increased disease self-management. However, eHealth interventions are often static and thereby less effective, and also frequently developed without (sufficiently) engaging end-users. Involving end-users, including those from lower SEP groups, and other relevant stakeholders can help to optimize the adoption and adherence to the eHealth intervention and result in the maintenance of healthy behavior.

The Perfect Fit intervention is the result of interdisciplinary collaboration, and the personalized eHealth intervention supports adult smokers to stop smoking and increase their PA using a virtual coach. We primarily aim to examine the feasibility, acceptability and preliminary effectiveness of the Perfect Fit intervention.

A mixed-method single-arm pre-post intervention study will be used. The intervention, delivered through a virtual coach, has a personalized duration and intensity, but will last on average 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Current smoker (cigarette, cigar, or rolling tobacco)
* Intention to quit smoking between now and 6 weeks
* Being able to walk without pain complaints
* Being able to understand and read Dutch (B1 level)
* Having access to the internet and a smartphone

In addition, at least 50% of sample has ≥10% risk of CVD (Nederlands Huisartsen Genootschap, 2019), estimated on basis of:

- Being female and 55+ years old OR male and 50+ years old

Finally, at least 75% of sample is:

- Living in region Leiden (region between Leiden/Amsterdam/Utrecht)

Exclusion Criteria:

* Being involved in smoking cessation therapy/counseling at the start of the intervention.
* Has undergone major lower extremity surgery in the past year (to prevent giving PA advice that contradicts medical guidance).
* Taking antipsychotics or having a serious psychiatric illness (e.g., schizophrenia/psychosis, bipolar disorder, major depression).
* Being pregnant.
* Not able to wear the smartwatch throughout the day (e.g., when individuals are not allowed to wear a watch at work)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Perfect Fit intervention assessed by completed intervention components and frequency of contact with the coach | Assessed after the intervention, at week 16 (post-intervention, T1)
  Assess feasibility of the Perfect Fit intervention using:
  1. usage data on which components of the intervention (i.e., chat conversations, exercises, informational videos) are completed at certain timepoints (measured from baseline to post-intervention, T1). Users who complete all the preparation phase dialogs, complete at least one dialog per week during the execution phase of the intervention, and complete the closing dialogue, will be marked as adherent users.
  2. a self-report question about the frequency of contact with the virtual coach; Users will be asked to indicate how many times a week they had contact with their virtual coach during the Perfect Fit intervention.
Acceptability of the Perfect Fit intervention assessed by the CSQ-8 | Assessed after the intervention, at week 16 (post-intervention, T1)
  Participants' satisfaction with the Perfect Fit intervention and the chat function of the NiceDay app (the app that is used for chat interaction between the user and the virtual coach) will be measured with the Dutch translation of the 8-item Client Satisfaction Questionnaire (CSQ-8; De Wilde & Hendriks, 2005; Larsen, 1979). An example of an item is: "To what extent has our service [the Perfect Fit program] met your needs?". The items are scored on 4-point Likert scales with different labels (e.g., from 1 (quite dissatisfied) to 4 (very satisfied)) and the total score ranges from 8 to 32, with a higher score indicating greater satisfaction.
Usability of the Perfect Fit intervention assessed by the SUS | Assessed after the intervention, at week 16 (post-intervention, T1)
  The usability of the Perfect Fit intervention and the chat function of the NiceDay app will be measured with a Dutch translation of the System Usability Scale (SUS; Brooke, 1996). The total questionnaire consists of ten items with items such as "I think the virtual coach is unnecessary complex" and "I found the various functions in this system were well integrated". The items are rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree).
Attitudes to the virtual coach assessed by satisfaction and relationship with, usability of and adherence to the virtual coach | Assessed after the intervention, at week 16 (post-intervention, T1)
  Acceptance of the virtual coach will be assessed using a Dutch translation of a set of six items that measure the evaluation of the coach in terms of satisfaction, usability, continuation of collaboration, relationship, preference for a program with or without coach and adherence to advice from the coach. The questionnaire has been used in other studies evaluating virtual agents (Bickmore et al., 2010; Provoost et al., 2020). Two example items are: "How satisfied were you with the virtual coach?" and "How easy was it talking to the virtual coach?". Answers are given on a 7-point Likert scale with different labels (e.g., from 1 (not at all satisfied) to 7 (very satisfied)).
Qualitative data on primary outcome measures | Assessed after the intervention, at week 16 (post-intervention, T1)
  Qualitative individual semi-structured interviews with participants will complement the quantitative data and provide more in-depth insight into acceptability, feasibility, preliminary effectiveness, and requirements for implementation of the Perfect Fit intervention.

SECONDARY OUTCOMES:
Preliminary effectiveness of the Perfect Fit intervention: Self-reported smoking abstinence | Assessed four times during the study: at post-intervention (week 16, T1), 2-month follow-up (week 24, T2), 6-month follow-up (week 40, T3), and 12-month follow-up (week 64, T4).
  To assess prolonged smoking abstinence at multiple timepoints after the Perfect Fit intervention, a combination of continuous abstinence and 7-day point prevalence abstinence will be used (Secades-Villa et al., 2016; Velicer & Prochaska, 2004; West et al., 2005). Participants will be asked if they have smoked since the end of the Perfect Fit intervention (yes/no; i.e., continuous abstinence). In case their answer is 'yes', participants will be asked if they have smoked the seven days prior to the assessment (yes/no; i.e., 7-day point prevalence abstinence). In case their answer to this question is 'no', two other follow-up questions will be asked, namely: "How long ago did you smoke your last cigarette, cigar or rolling tobacco?" and "How many cigarettes, cigars or rolling tobacco did you smoke?'.
Preliminary effectiveness of the Perfect Fit intervention: Self-reported level of PA | Assessed five times during the study: at baseline (week 0, T0), post-intervention (week 16, T1), 2-month follow-up (week 24, T2), 6-month follow-up (week 40, T3), and 12-month follow-up (week 64, T4).
  Self-reported level of PA will be measured with a Dutch translation of the 3-item Godin-Shephard Leisure-Time PA questionnaire (GSLTPAQ; Amireault & Godin, 2015; Godin, 2011). Participants are asked how many times on average, during a typical week, they do strenuous, moderate or mild exercise for more than 15 minutes. The total score of the questionnaire is calculated by multiplying the number of times per week strenuous exercise by nine, multiplying the number of times per week moderate exercise by five, multiplying the number of times per week mild exercise by three, and taking the sum of this (i.e., (9 x times/wk strenuous) + (5 x times/wk moderate) + (3 x times/wk mild)). A total score of 24 or more is defined as 'active', a total score of 14 to 23 is defined as 'moderately active' and a score of less than 14 is defined as 'insufficiently active' (Godin, 2011).
Preliminary effectiveness of the Perfect Fit intervention: non-smoker self-identity | Assessed five times during the study: at baseline (week 0, T0), post-intervention (week 16, T1), 2-month follow-up (week 24, T2), 6-month follow-up (week 40, T3), and 12-month follow-up (week 64, T4).
  Non-smoker self-identity will be assessed using seven items (Meijer et al., 2016), of which three are adapted from the Abstainer Self-Concept scale and three are adapted from the Smoker Self-Concept Scale (Shadel & Mermelstein, 1996) by replacing 'smoking' with 'not smoking'. In addition, the item "I would like to be a non-smoker" will be added (adapted from Tombor et al., 2013). All items are translated to Dutch and can be answered on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Higher total scores indicate stronger non-smoker self-identity.
Preliminary effectiveness of the Perfect Fit intervention: PA self-identity | Assessed five times during the study: at baseline (week 0, T0), post-intervention (week 16, T1), 2-month follow-up (week 24, T2), 6-month follow-up (week 40, T3), and 12-month follow-up (week 64, T4).
  PA self-identity will be measured with a Dutch translation of the adapted version (Strachan et al., 2010) of the 9-item Exercise Identity Questionnaire (Anderson & Cychosz, 1994). PA identity will be measured rather than exercise identity since being physically active entails a broader array of physical activities (Strachan et al., 2010). As the Perfect Fit intervention aims to enhance PA by increasing the amount of steps, this includes not only sports/exercise, but also daily physical activities like household chores. An example item is: "I consider myself a physically active person". Answers are given on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree) and the total score ranges from 9 to 63, with a higher score indicating stronger identity.
Preliminary effectiveness of the Perfect Fit intervention: Smoking abstinence self-efficacy | Assessed five times during the study: at baseline (week 0, T0), post-intervention (week 16, T1), 2-month follow-up (week 24, T2), 6-month follow-up (week 40, T3), and 12-month follow-up (week 64, T4).
  Smoking abstinence self-efficacy will be assessed with a single item (adapted from Loprinzi et al., 2015), translated in Dutch. Participants will be asked: "Overall, how confident are you that you are able not to smoke ?". Abstinence self-efficacy has been shown to be associated with smoking cessation (Spek et al., 2013). Answers are given on a 5-point Likert scale ranging from 1 (not at all confident) to 5 (extremely confident), with a higher score indicating higher abstinence self-efficacy.
Preliminary effectiveness of the Perfect Fit intervention: PA self-efficacy | Assessed five times during the study: at baseline (week 0, T0), post-intervention (week 16, T1), 2-month follow-up (week 24, T2), 6-month follow-up (week 40, T3), and 12-month follow-up (week 64, T4).
  To assess self-efficacy for PA the same Dutch single item (adapted from Loprinzi et al., 2015) will be used as for assessing smoking abstinence self-efficacy, but the item will be adjusted to PA behavior: "Overall, how confident are you that you are able to be sufficiently physically active?". An instruction will be provided before the question is presented, explaining the definition of PA (i.e., exercise, but also physical activities like walking to the supermarket) and the recommended levels of PA according to the WHO guidelines (World Health Organisation, 2022). PA self-efficacy has been shown to be associated with actual PA behavior (McAuley & Blissmer, 2000). Answers are given on a 5-point Likert scale ranging from 1 (not at all confident) to 5 (extremely confident), with a higher score indicating higher self-efficacy for PA.
Preliminary effectiveness of the Perfect Fit intervention: Objective level of PA | Assessed during the intervention: from baseline (week 0, T0) to post-intervention (week 16, T1)
  The average number of steps per day will be measured with the smartwatch participants are wearing during the study and collected using the sensor data collector app. The sensor data will be collected during the Perfect Fit intervention.
Feasibility of the study: Recruitment, response and consent rate | Assessed from the start of the recruitment till inclusion of final participant
  Feasibility of the study will be assessed in terms of recruitment, response and consent rate using participant screening and inclusion logfile data. The following information will be logged: the time between the start of patient recruitment and the day on which the final participant is recruited (i.e., recruitment rate); proportion of interested participants who completed screening questionnaire (i.e., response rate); and number of eligible participants who consented to take part in study (i.e., consent rate).
Feasibility of the study: Recruitment strategies | Assessed before the intervention, at baseline (week 0, T0)
  To gain more insight in the effectiveness of different recruitment strategies, participants will be asked at baseline how they heard about the study. They can indicate which recruitment strategy was used (e.g., recruited directly by a researcher, via social media post). This will provide insight in effective recruitment strategies for future research, which is especially interesting in the case of participants with a lower SEP as they are often underrepresented in research.
Feasibility of the study: Adherence | Assessed from the start of the recruitment to the end (week 64, T4) of the study
  Users' adherence to the study will be assessed using participant log data. Adherence will be examined in terms of the number of participants who completed the Perfect Fit intervention and the study, the number of participants lost to follow-up over time (dropouts), and the number of participants who do not drop out from the study, i.e. still filling in questionnaires, but who are no longer using the app (nonusers; Eysenbach, 2005). Adherence will be monitored during the full study duration by keeping a participant screening and inclusion logfile and will also be assessed with the earlier mentioned usage data and self-report question (see primary outcome 'Feasibility of the Perfect Fit intervention').
Feasibility of the study: Intervention completion after 16 weeks | Assessed after the intervention, at week 16 (post-intervention, T1)
  At the start of the post-intervention questionnaire, users will be asked if they completed the intervention (i.e., completed the final closing dialog with the virtual coach) or not. In case they did not complete the intervention yet, they are asked in which week of the execution phase of the Perfect Fit intervention they are at that moment. This way it can be assessed if participants fill out the post-intervention questionnaire while having completed the whole intervention or not. It also provides information on how many people complete the intervention in 16 weeks or less.
Qualitative data on secondary outcome measures | Assessed after the intervention, at week 16 (post-intervention, T1)
  Qualitative individual semi-structured interviews with participants will complement the quantitative data and provide more in-depth insight into acceptability, feasibility, preliminary effectiveness, and requirements for implementation of the Perfect Fit intervention.

OTHER OUTCOMES:
Demographic characteristics | Assessed before the intervention, at baseline (week 0, T0)
  General information about the participants will be obtained, namely gender (i.e., male, female, other), age (birth year), level of education (i.e., primary education, vmbo, havo, vwo, mbo, hbo, wo; as measure for SEP), if they currently have any physical or psychiatric/mental (chronic) condition(s) and eHealth literacy. To assess eHealth literacy a validated Dutch translation (Poot et al., 2023) of the eHealth Literacy Questionnaire (eHLQ) will be used (Kayser et al., 2018). Five of the seven dimensions will be used: 1) Using technology to process health information; 2) Understanding of health concepts and language; 3) Ability to actively engage with digital services; 4) Feel safe and in control; and 5) Motivated to engage with digital services. Each dimension consists of five items, resulting in 25 items in total. Each item is scored on a 4-point scale (strongly disagree (1), disagree (2), agree (3), strongly agree (4)), with a higher score indicating higher eHealth literacy.
Intention to quit smoking | Assessed before the intervention, at baseline (week 0, T0)
  Participants will be asked for an intended timeline to quit smoking in the future. Answer categories are based on the stages of change of the Transtheoretical model (Prochaska & DiClemente, 2005) and include: within the next month (1), between 1 to 6 months from now (2), sometime in the future, beyond 6 months (3) or not planning to quit (4; Hummel et al., 2018). Participants who choose answer category four will be categorized as 'non-intenders'. This variable will be recoded so that higher scores indicate stronger intention to quit. Since intention to quit smoking is also one of the inclusion criteria, we expect that participants in the study are not likely to choose answer option 3 and 4.
Physical nicotine dependence | Assessed before the intervention, at baseline (week 0, T0)
  Physical nicotine dependence will be assessed using the Dutch version of the Fagerström Test of Nicotine Dependence (FTND; Heatherton et al., 1991; Penfornis et al., 2021). The FTND consists of six items, of which four items are scored on a dichotomous scale (yes / no), one item is scored using four answer categories, and one item has an open answer format (asking participants about the number of cigarettes smoked per day). An example item is "Do you smoke more in the morning than during the rest of the day?". Total scores can range from 5 to 12, with a higher score indicating higher nicotine dependence.
Intention to become more physically active | Assessed before the intervention, at baseline (week 0, T0)
  The same question is used as for intention to quit smoking. First, an instruction will be provided before the question is presented, explaining the definition of PA (i.e., exercise, but also physical activities like walking to the supermarket) and the recommended levels of PA according to the WHO guidelines (World Health Organisation, 2022). Then participants are asked to indicate whether they intend to become more physically active. Answer categories are based on the stages of change of the Transtheoretical model (Prochaska & DiClemente, 2005) and include: within the next month (1), between 1 to 6 months from now (2), sometime in the future, beyond 6 months (3) or not planning to become more physically active (4; Hummel et al., 2018). Participants who choose answer category four will be categorized as 'non-intenders'. This variable will be recoded so that higher scores indicate stronger intention to become more physically active.
Use of additional aids/support for smoking cessation or PA enhancement | Assessed four times during the study: at post-intervention (week 16, T1), 2-month follow-up (week 24, T2), 6-month follow-up (week 40, T3), and 12-month follow-up (week 64, T4).
  Participants will be asked if they made use of additional aids or support for smoking cessation or PA enhancement. Participants are asked if they have used any type of additional support (e.g., medication, booklets, websites, other apps, or treatment/support, like professional coaching, a sport challenge or acupuncture) next to the Perfect Fit intervention, and if so, what type of support. This will provide insight in other forms of support that were used and could influence the results. It will also provide insight in the applicability of the intervention (e.g., use as stand-alone or add-on intervention).
Self-reported (re)lapses during intervention after quit date | Assessed during the intervention, from the moment the quit date is set (around week 2-4) till post-intervention (week 16, T1)
  Lapses (defined as one time point of smoking again after the quit date, any quantity) and relapses (defined as multiple time points of smoking again after the quit date, any quantity) during the execution phase (i.e., phase which starts on the quit date) of the Perfect Fit intervention will be assessed using usage data. Usage data about cigarettes smoked after the quit date will be obtained in two ways. First, as part of the '(re)lapse dialog' with the coach. This dialog can be initiated by the user in case of (re)lapse to receive support from the coach to cope with this (re)lapse. During this dialog the coach will ask the user if it concerns a lapse or a relapse and how many cigarettes they smoked. Second, via the 'tracker' functionality of the NiceDay app. Users can use this functionality during the whole Perfect Fit intervention. Both ways of obtaining data on (re)lapses rely on self-report of the user.
Smoking e-cigarettes | Assessed five times during the study: at baseline (week 0, T0), post-intervention (week 16, T1), 2-month follow-up (week 24, T2), 6-month follow-up (week 40, T3), and 12-month follow-up (week 64, T4).
  Participants will also be asked if they smoke/use e-cigarettes. In case their answer to this question is 'yes', they will be asked if they smoke e-cigarettes with or without nicotine and how often. This is assessed as some people switch to e-cigarettes after quitting smoking tobacco.
Self-reported level of occupational PA | Assessed five times during the study: at baseline (week 0, T0), post-intervention (week 16, T1), 2-month follow-up (week 24, T2), 6-month follow-up (week 40, T3), and 12-month follow-up (week 64, T4).
  Since the level of PA during work can differ between participants, participants will also be asked about the level of PA during their workday using a single item: "How would you describe your daily physical activity at work? Choose the answer that best suits your work activities:". The answer options are partly based on the Occupational Sitting and Physical Activity Questionnaire (OSPAQ; Reis et al., 2005) and the Global Physical Activity Questionnaire (GPAQ; Armstrong & Bull, 2006) and include: 1) Mostly sedentary (I sit almost all day and do little or no physical activity), 2) mild exercise (I am involved in light physical activities such as standing and occasionally walking, but not intensively), 3) moderate intensity exercise (I perform activities that require moderate physical exertion, such as fast walking, lifting light loads), 4) strenuous exercise (I mainly engage in physically demanding activities, such as heavy lifting), or 5) I am not working at the moment.

CONTACTS AND LOCATIONS:
Overall Officials: Anke Versluis, Dr., Principal Investigator — Leiden University Medical Center (LUMC); Eline Meijer, Dr., Principal Investigator — Leiden University Medical Center (LUMC)
Locations (1):
- Leiden University Medical Center (LUMC), Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized data will be made available for reuse at the end of the project. Certain demographic characteristics might have to be removed from the data set, to prevent traceability of individual participants. It has yet to be decided whether data can best be made available through a repository or through reasonable request.
Supporting Information: Study Protocol